CLINICAL TRIAL: NCT07194915
Title: Pleural Fluid Neutrophil Extracellular Traps Exacerbate Disease Severity and Risk of One-year Mortality in Pleural Infection: An Observational, International, Multicohort Study (TORPIDS-3)
Brief Title: Pleural Fluid Neutrophil Extracellular Traps Exacerbate Disease Severity and Risk of One-year Mortality in Pleural Infection (TORPIDS-3)
Acronym: TORPIDS-3
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: TORPIDS-3
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Pleural Infection
Keywords: pleural infection; neutrophils; neutrophil extracellular traps; NETs; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Acellular pleural fluid specimens were analysed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- PILOT: Pleural fluid specimens collected for the PILOT study
- Oxford Pleural Biobank: Pleural fluid specimens collected in Oxford
- Oxford-Osler: Pleural fluid specimens collected in Oxford
- Patras Pleural Biobank: Pleural fluid specimens collected in Patras, Greece
- Ancona Pleural Biobank: Pleural fluid specimens collected in Ancona, Italy

SUMMARY:
Pleural infection is a severe and complicated disease which is associated with significant morbidity and mortality. People with pleural infection show diverse levels of neutrophil degranulation activity. The investigators examined the biological role of pleural fluid neutrophil extracellular traps in patients with pleural infection. TORPIDS-3 is an observational, International multicohort study.

ELIGIBILITY:
Inclusion Criteria:

Patients were included if they had a clinical presentation consistent with pleural infection as stated in the Methods section of the main manuscript and any of the following criteria:

1. Pleural fluid that was macroscopically purulent, OR
2. Pleural fluid that was positive on culture for bacterial infection, OR
3. Pleural fluid that demonstrated bacteria on Gram staining, OR
4. Pleural fluid with pH ≤7.2 (measured in a blood gas analyser) or low glucose level (≤3mmol/L or ≤55mg/dL) in a patient with clinical evidence of infection, OR
5. Contrast-enhanced CT evidence of pleural infection (consolidation of underlying lung with enhancing pleural collection) in a patient with clinical evidence of infection, alongside exclusion of other sources of infection.

Exclusion criteria:

1. Age less than 18 years, OR
2. No pleural fluid available for analysis, OR
3. Patient previous pneumonectomy on the side of pleural infection, OR
4. Expected survival less than three months due to co-morbid disease, as judged by the recruiting physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed pleural infection
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Disease severity | Baseline
  Association between pleural fluid NETs with disease severity
One-year mortality | Baseline
  Association between pleural fluid NETs and risk of one-year mortality

SECONDARY OUTCOMES:
Bacterial profiles | Baseline
  Association between pleural fluid NETs with bacterial profiles
Sonographic septations | Baseline
  Association between pleural fluid NETs and the presence of sonographic septations
Need for Intrapleural Enzyme Therapy (IET) | Baseline
  Association between pleural fluid NETs with the requirement for IET

CONTACTS AND LOCATIONS:
Locations (1):
- CAMS Oxford Institute, Nuffield Department of Medicine, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corcoran JP, Psallidas I, Gerry S, Piccolo F, Koegelenberg CF, Saba T, Daneshvar C, Fairbairn I, Heinink R, West A, Stanton AE, Holme J, Kastelik JA, Steer H, Downer NJ, Haris M, Baker EH, Everett CF, Pepperell J, Bewick T, Yarmus L, Maldonado F, Khan B, Hart-Thomas A, Hands G, Warwick G, De Fonseka D, Hassan M, Munavvar M, Guhan A, Shahidi M, Pogson Z, Dowson L, Popowicz ND, Saba J, Ward NR, Hallifax RJ, Dobson M, Shaw R, Hedley EL, Sabia A, Robinson B, Collins GS, Davies HE, Yu LM, Miller RF, Maskell NA, Rahman NM. Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study. Eur Respir J. 2020 Nov 26;56(5):2000130. doi: 10.1183/13993003.00130-2020. Print 2020 Nov. PMID 32675200